CLINICAL TRIAL: NCT03413488
Title: Kinesio Taping Compared to Exercise Intervention for Round Shoulder Subjects With Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201705117RIND
Record Dates: First submitted 2018-01-11; First posted 2018-01-29 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-02

CONDITIONS: Shoulder Impingement Syndrome (SIS); Round Shoulder Posture (RSP)
Keywords: Shoulder impingement syndrome; Kinesio tape; Round shoulder posture
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping (Experimental): subject with shoulder impingement syndrome
  Interventions: Other: kinesio taping
- Exercise (Active Comparator): subject with shoulder impingement syndrome
  Interventions: Other: exercise

INTERVENTIONS:
Other: kinesio taping — Apply exercise and kinesio taping for intervention
  Arms: Kinesio taping
Other: exercise — Apply only exercise intervention
  Arms: Exercise

SUMMARY:
To compare the effect between the exercise intervention (strengthening exercise and stretching exercise) and exercise intervention with taping on decreasing round shoulder posture and improving symptoms in subjects with shoulder impingement syndrome/round shoulder syndrome.

DETAILED DESCRIPTION:
Background: Poor posture and abnormal scapular kinematics have been suggested as possible primary factors in developing Shoulder impingement syndrome (SIS) and also as secondary observed phenomena of SIS. Round shoulder posture (RSP) is major and common posture contributing to increase the potential for subacromial impingement or exaggerate the symptoms of SIS. Objective: To compare the effect between the exercise intervention (strengthening exercise and stretching exercise) and exercise intervention with taping on decreasing RSP and improving symptoms in subjects with SIS/RSP. Methods: Forty subjects with impingement age between 20 and 75 are recruited and measured on acromial distance, pectoralis minor index (PMI), posterior and anterior shoulder tightness, distance of scapular medial border, pain score and flexilevel scale of shoulder function (FLEX-SF). Clinical significance: Shoulder impingement syndrome (SIS) have been identified as the majority of reported shoulder complaints. The project will provide an effective intervention for subjects with SIS/RSP.

ELIGIBILITY:
Inclusion criteria:

1. subjects age between 20 and 75
2. Diagnosed with shoulder impingement syndrome
3. At least three positive of five tests, including Neer's test, Hawkin's test, Empty can test, tenderness in tendon of rotator cuff

Exclusion criteria:

1. Shoulder pain onset due to trauma
2. A history of shoulder fractures or dislocation
3. Cervical radiculopathy
4. Degenerative joint disease of the shoulder
5. Surgical interventions on the shoulder
6. Inflammatory arthropathy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Length of the pectoralis minor | 1 year
  The Pectoralis minor index (PMI) is calculated by dividing the resting muscle length by the subject's height and multiplying by 100.
Acromial distance (AD) | 1 year
  Acromial distance is defined as the distance from table to border of lateral-inferior acromion and measured in centimeter.
Posterior and anterior shoulder tightness | 1 year
  Flexibility of the posterior and anterior shoulder tissues, measured in degree
Distance of scapular medial border | 1 year
  The distance from the root of the spine (ROS) and the inferior angle (INF) of the scapula to the thoracic wall in millimeter respectively
Self-reported flexilevel scale of shoulder function (FLEX-SF) | 1 year
  FLEX-SF is used to assess shoulder function and disability. Scores will be recorded from 1, with the most limited function, to 50, without any limited function in the subject.
Pain score | 1 year
  Severity of pain is measured by Visual Analogue Scale, providing a range of scores from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Lan Yang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan